CLINICAL TRIAL: NCT06226909
Title: The Efficacy of Shear-wave Elastography-guided Biopsy for Diagnosis in Pleural Disease: a Randomized Controlled Trial
Brief Title: The Efficacy of Shear-wave Elastography-guided Biopsy for Diagnosis in Pleural Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 202311139RINC
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Pleural Diseases
MeSH Terms: conditions — Pleural Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shear-wave elastography-guided (Experimental): based on the shear-wave elastography, the area with the highest elasticity value will be the target area to perform pleural biopsy for at least 6 times
  Interventions: Procedure: different types of ultrasound technique
- B-mode ultrasound-guided (Active Comparator): based on the B-mode transthoracic ultrasound, the area with the maximal thickness will be the target area to perform pleural biopsy for at least 6 times
  Interventions: Procedure: different types of ultrasound technique

INTERVENTIONS:
Procedure: different types of ultrasound technique — Shear-wave elastography-guided or B-mode ultrasound-guided

SUMMARY:
To investigate the information from shear-wave elastography on pleural tissues will improve the diagnosis of pleural diseases, as to increase the diagnostic yield in ultrasound-guided transthoracic pleura biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with radiographic evidence of pleural disease

Exclusion Criteria:

* Age < 18 y/o
* Patients who cannot hold their breath for 5 seconds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
The diagnostic yield of the two groups | 6 months
  the pathology of pleural biopsies will be interpreted by cytopathologists

SECONDARY OUTCOMES:
Procedure time | 1 day
  Procedure time
the rate of pneumothorax & hemothorax | 1 day
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Yao-Wen Kuo, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No